CLINICAL TRIAL: NCT03323463
Title: A Prospective Single Arm Non-inferiority Trial of Major Radiation Dose De-Escalation Concurrent With Chemotherapy for Human Papilloma Virus Associated Oropharyngeal Carcinoma (Major De-escalation to 30Gy for Select Human Papillomavirus Associated Oropharyngeal Carcinoma)
Brief Title: Major De-escalation to 30 Gy for Select Human Papillomavirus Associated Oropharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-409
Record Dates: First submitted 2017-10-17; First posted 2017-10-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HPV-Associated Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Neck
Keywords: squamous cell carcinoma of the neck of unknown primary; HPV-Associated Oropharyngeal Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; 17-409; Hypoxia negative; N1-2c oropharyngeal squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Carboplatin; Fluorouracil; Proton Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm A: HPV associated oropharyngeal carcinoma (Experimental): HPV associated oropharyngeal carcinoma subjects who also have no evidence of hypoxia. This arm is closed to accrual.
  Interventions: Diagnostic Test: F-FMISO PET/CT Scan; Radiation: 30 Gy over 3 weeks; Drug: Cisplatin; Drug: Carboplatin; Drug: 5Fluorouracil
- Arm B: HPV associated oropharyngeal carcinoma (Experimental): HPV associated oropharyngeal carcinoma subjects who also have no evidence of hypoxia.
  Interventions: Diagnostic Test: F-FMISO PET/CT Scan; Radiation: 30 Gy over 3 weeks; Drug: Cisplatin; Drug: Carboplatin; Drug: 5Fluorouracil; Radiation: Proton Therapy

INTERVENTIONS:
Diagnostic Test: F-FMISO PET/CT Scan — All subjects on Cohort A and the first 100 subjects accrued to Cohort B will undergo a pre-treatment F-FMISO scan PET/CT scan pretreatment. For both Cohort A and Cohort B, FMISO scan will be repeated between the 5th-10th RT day if pre-treatment scan is hypoxic. If the repeat 18F-FMISOscan PET/CT demonstrates hypoxia, the subject will receive 70Gy concurrent with 2 cycles of chemotherapy. All subjects accrued onto Cohort B after 100 accruals will undergo only one 18F-FMISO scan done 5-10 treatment days after start of radiation therapy.
Radiation: 30 Gy over 3 weeks — Treatment will be delivered as one fraction per day on a standard 5 day per week schedule (excluding weekends and holidays), total of 30 Gy over 3 weeks at 2 Gy per fraction each day. The gross nodes, the primary/postoperative bed if applicable, all subclinical areas at risk for disease will receive the same dose at 30Gy.
Drug: Cisplatin — Cycle 1 (week 1): At the start of week 1 of IMRT, subjects will receive cisplatin 100 mg/m2 intravenously. They may be given for 2 consecutive days (50 mg/m2 each day for a total dose 100 mg/m2), typically on days 1 and 2, or as a single dose, typically on day 1.
Drug: Carboplatin — If cisplatin cannot be given at 100 mg/m2 for either cycle 1 or cycle 2, the investigator may use a regimen with carboplatin and 5-Fluorouracil in its place. Carboplatin will be given at a dose of AUC 1.25 intravenously daily x 4 days starting on day 1 of the cycle (total dose of AUC 5). Cycle 2 (Week 4): After the three weeks of radiation at week 4 when the subject no longer is receiving radiation therapy, subjects will receive cisplatin 100 mg/m2 intravenously. The may be given for 2 consecutive days (50 mg/m2 each day for a total dose 100 mg/m2), typically on days 22 and 23, or as a single dose, typically on day 22.
Drug: 5Fluorouracil — If cisplatin cannot be given at 100 mg/m2 for either cycle 1 or cycle 2, the investigator may use a regimen with carboplatin and 5-Fluorouracil in its place. 5-Fluorouracil will be given at a dose of 600 mg/m2 intravenous infusion over 24 hours daily x 4 days (total dose of 2400 mg/m2 intravenous infusion over 96 hours).
Radiation: Proton Therapy — Proton beam using pencil beam delivery either with the Varian or IBA delivery systems will be allowed for Cohort B. Proton beam therapy will be given at the New York Proton Center in New York City, where MSKCC has a well-established business associate agreement and cooperative research agreement with, respectively. If treatment at NYPC is not feasible, patients may be referred to ProCure in Somerset, NJ.
  Arms: Arm B: HPV associated oropharyngeal carcinoma

SUMMARY:
The purpose of this study is to demonstrate that participants with HPV positive and hypoxia negative T1-2, N1-2c (AJCC, 7th ed.) oropharyngeal squamous cell carcinoma receiving a major de-escalated radiation therapy with 2 cycles of standard chemotherapy is not inferior to comparable subjects treated with the current standard chemoradiation.

Accrual for Cohort A has been completed.

Cohort B is active and continues to enroll participants where surgery is optional and proton is allowed.

DETAILED DESCRIPTION:
This non-randomized non-inferiority study will enroll HPV associated oropharyngeal carcinoma subjects. Subjects who also have no evidence of hypoxia will undergo a major de-escalated radiation therapy concurrent with standard chemotherapy. Hypoxia status will be determined by 1 BF-FMISO PET /CT imaging. If this baseline scan shows no evidence of hypoxia, the subject will receive 30Gy concurrent with 2 cycles of chemotherapy. If this baseline scan shows evidence of hypoxia, a repeat 1 BF-FMISO scan will be done 5-10 treatment days after start of radiation therapy. If the repeat 1 BF-FMISO scan PET /CT demonstrates no evidence of hypoxia, the subject will receive 30Gy concurrent with 2 cycles of chemotherapy. If the repeat 1 BF-FMISO scan PET /CT demonstrates hypoxia, the subject will receive 70Gy concurrent with 2 cycles of chemotherapy. At 4 (+/- 4 weeks) months after chemoradiation, a neck dissection will be done unless the subjects FDG PET /CT scan at that time shows no evidence of disease of which the subject can be observed as per current standard of care.

ELIGIBILITY:
Inclusion Criteria:

- Cohort A: Pathologically (histologically or cytologically) proven diagnosis of HPV associated squamous cell carcinoma of the oropharynx (tonsil, base of tongue, or oropharyngeal walls) from surgical resection or excisional biopsy regardless of margin status.

* Squamous cell carcinoma of the neck of unknown primary is allowed with excision biopsy of a lymph node (or core biopsy) and consent from the PI or co-PIs

  * Cohort B: Pathologically (histologically or cytologically) proven diagnosis of HPV associated squamous cell carcinoma of the oropharynx (tonsil, base of tongue, or oropharyngeal walls). Surgical removal of primary site is no longer required.
* Squamous cell carcinoma of the neck of unknown primary is allowed with excision biopsy of a lymph node (or core biopsy) and consent from the PI or co-PIs

  * Subjects must have clinically or radiographically evident measurable disease at nodal stations.
  * Clinical stage T1-2, N1-2c without evidence of distant metastasis based on FDG PET/CT.
* Patients who have squamous cell carcinoma of the neck of unknown primary, and thus, are T0, are allowed with excision biopsy of a lymph node (or core biopsy) or consent from the PI or co-PI

  * CT or MRI of the neck with and without contrast Note: A CT scan of neck and/or a PET/CT performed for the purposes of radiation planning may serve as planning tools.
  * ECOG Performance Status of 0-2 or Karnopsky Performance Status >/= 50
  * Age ≥ 18
  * Adequate hematologic function within 30 days prior to registration, defined as follows:
* White Blood Count (WBC) >/= 2 K/mcL
* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
* Platelets ≥ 100,000 cells/mm3
* Hemoglobin ≥ 8.0 g/dl; Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable

  * Adequate renal function within 30 days prior to registration, defined as follows:
* Serum creatinine ≤ 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula

CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)

* Adequate hepatic function within 30 days prior to registration, defined as follows:

  * Bilirubin ≤ 2 mg/dl
  * AST or ALT ≤ 3 x the upper limit of normal
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential
* The subject must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Subjects with prior head and neck radiation therapy
* Subjects with simultaneous primary cancers outside of the oropharynx
* Note: Exceptions can be made for patients with simultaneous primaries outside the oropharynx if determined by the PI/Co-PI the patient can proceed with protocol activities
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for 3 years or if cure rate from treatment at 5 years to be 90% or greater
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* No particle therapy such as but not limited to proton therapy is allowed in Cohort A. For Cohort B, this exclusion is removed.
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  * Hepatic Insufficiency resulting in clinical jaundice and/or coagulation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of study treatment for participants receiving de-escalated radiation therapy radiation therapy, comparable to participants treated with the current standard of care chemoradiation by standard CT (or MRI) or tumor site and PET scan | 2 years (+/- 3 months)
  The primary objective of this protocol is to demonstrate that the 2-year locoregional control for this cohort of subjects treated with a major de-escalated radiation dose of 30 Gy is not inferior to comparable subjects treated with the current standard chemoradiation at 70 GY by using a proportion test of patients who demonstrate 2-year locoregional control.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Hartford Healthcare (Data Collection), Hartford, Connecticut
  - Baptist Alliance MCI (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee NY, Sherman EJ, Schoder H, Wray R, Boyle JO, Singh B, Grkovski M, Paudyal R, Cunningham L, Zhang Z, Hatzoglou V, Katabi N, Diplas BH, Han J, Imber BS, Pham K, Yu Y, Zakeri K, McBride SM, Kang JJ, Tsai CJ, Chen LC, Gelblum DY, Shah JP, Ganly I, Cohen MA, Cracchiolo JR, Morris LGT, Dunn LA, Michel LS, Fetten JV, Kripani A, Pfister DG, Ho AL, Shukla-Dave A, Humm JL, Powell SN, Li BT, Reis-Filho JS, Diaz LA, Wong RJ, Riaz N. Hypoxia-Directed Treatment of Human Papillomavirus-Related Oropharyngeal Carcinoma. J Clin Oncol. 2024 Mar 10;42(8):940-950. doi: 10.1200/JCO.23.01308. Epub 2024 Jan 19. PMID 38241600
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org